CLINICAL TRIAL: NCT01153542
Title: An Open-Label Phase 1 Study to Examine the Effect of VX 770 on Desipramine in Healthy Subjects
Brief Title: Study of VX-770 on Desipramine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Claudia Ordonez, MD, Vertex Pharmaceuticals, Inc.
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VX10-770-011
Record Dates: First submitted 2010-06-28; First posted 2010-06-30 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-12

CONDITIONS: In Development for Cystic Fibrosis
MeSH Terms: interventions — ivacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VX-770 (Experimental)
  Interventions: Drug: VX-770
- desipramine (Experimental)
  Interventions: Drug: VX-770

INTERVENTIONS:
Drug: VX-770 — In period 1, subjects will receive a single oral dose of desipramine on Day 1.
  Arms: desipramine
Drug: VX-770 — In period 2, subjects will receive 150 mg VX-770 q12h orally from the morning of Day 1 through the evening of Day 9. Subjects will receive 50 mg Desipramine as a single dose on Day 5 of period 2.

SUMMARY:
The objective of this study is to evaluate the effects of VX-770 on Desipramine

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be male or female and between 18 and 55 years of age
* Subject must have a body mass index (BMI) from 18 to 30 kg/m2
* Subject must be judged to be in good health

Exclusion Criteria:

* History of any illness that, in the opinion of the investigator or the subject's general practitioner, might confound the results of the study or pose an additional risk in administering study drug(s) to the subject
* Subjects who have human immunodeficiency virus, hepatitis C, or active hepatitis B
* Female subjects and male subjects with female partner(s) who are pregnant, nursing, or planning to become pregnant during the study or within 90 days of the last dose of study drug

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
VX-770 and Desipramine pharmacokinetic parameters | 3 weeks

SECONDARY OUTCOMES:
Safety as measured by adverse events, vital signs, electrocardiograms (ECGs), and clinically significant laboratory assessments | 3 weeks
Metabolites pharmacokinetic parameters in plasma | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: H. Frank Farmer, MD, Principal Investigator — Covance CRU, Inc.
Locations (1):
- Covance CRU, Inc., Daytona Beach, Florida, United States